CLINICAL TRIAL: NCT06055439
Title: A Phase 1/2 Study to Evaluate CHM-2101, an Autologous Cadherin 17 (CDH17) Chimeric Antigen Receptor (CAR) T Cell Therapy for the Treatment of Relapsed or Refractory Gastrointestinal Cancers
Brief Title: A Phase 1/2 Study to Evaluate CHM-2101, an Autologous Cadherin 17 Chimeric Antigen Receptor (CAR) T Cell Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chimeric Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHM-2101-001
Record Dates: First submitted 2023-09-13; First posted 2023-09-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Neuroendocrine Tumors; Colorectal Cancer; Gastric Cancer
MeSH Terms: conditions — Neuroendocrine Tumors; Colorectal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous CDH17 CAR T-cell Therapy (Experimental): After receiving three daily doses of IV fludarabine and cyclophosphamide, participants will receive a single dose of IV CHM-2101.
  The dose of CHM-2101 during Phase 1 will be based on "3+3" rules of dose escalation.
  The recommended Phase 2 dose will be based on results from the Phase 1.
  Interventions: Biological: CHM-2101 CAR-T cells

INTERVENTIONS:
Biological: CHM-2101 CAR-T cells — Cadherin 17 (CDH17) Chimeric Antigen Receptor (CAR)-positive T cells

SUMMARY:
The goal of this clinical trial is to evaluate CHM-2101, an autologous CDH17 CAR T-cell therapy for the treatment of advanced gastrointestinal (GI) cancers that are relapsed or refractory to at least 1 standard treatment regimen in the metastatic or locally advanced setting.

DETAILED DESCRIPTION:
This is a Phase 1/2 open-label study to evaluate CHM-2101, an autologous CDH17 CAR T-cell therapy for the treatment of advanced gastrointestinal (GI) cancers that are relapsed or refractory to at least 1 standard treatment regimen in the metastatic or locally advanced setting.

The study has 2 parts: Phase 1, Dose Escalation and Expansion, and Phase 2. Potential participants will provide written consent and be screened for study eligibility prior to undergoing any screening procedures, including leukapheresis. Protocol-specified criteria must be met prior to the start of leukapheresis for collection of peripheral blood mononuclear cells (PBMCs). Eligible participants will undergo leukapheresis to collect PBMCs for product manufacturing, which comprises enrichment of T cells, lentiviral transduction, ex vivo expansion, and cryopreservation of the CHM-2101 cell product. Participants who have a leukapheresis or manufacturing failure may be permitted a second attempt at leukapheresis.

Bridging chemotherapy (treatment between the time of leukapheresis and first dose of lymphodepleting chemotherapy [LDC]) is permitted at the discretion of the investigator, if needed to maintain disease stability during CHM-2101 manufacturing time. Bridging chemotherapy is prohibited within the 2 weeks prior to leukapheresis and 2 weeks prior to planned CHM-2101 infusion. Specific criteria to proceed should be reviewed prior to leukapheresis, LDC, and CHM-2101 infusion. Participants will be followed in this study for 18 months or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Documented informed consent of the participant and/or legally authorized representative.
2. Confirmed histologic diagnosis of one of the following solid tumors of GI origin:

   1. Gastric adenocarcinoma Note: for gastric adenocarcinoma patients only, central laboratory confirmation of CDH17+ tumor expression is required.
   2. Colon and/or rectal adenocarcinoma
   3. G1, G2, and well-differentiated G3 neuroendocrine tumors of the midgut and hindgut (ileal, jejunal, cecal, distal colonic, or rectal; with ≤ 55% Ki67 expression)
3. Availability of unstained tumor tissue slides from archived tumor tissue or a new tumor biopsy, if medically feasible. Note: for gastric adenocarcinoma patients only, confirmation of CDH17+ is required prior to study inclusion.
4. Have received at least 1 prior line of systemic anti-cancer treatment in the locally advanced or metastatic setting, as defined by National Comprehensive Cancer Network (NCCN) guidelines. Participants must have received or declined FDA-approved and available treatment options, including targeted therapies for disease mutation or antigen expression status.
5. Age ≥ 18 years and ≤ 85 years.
6. For Phase 1 Dose Expansion and Phase 2 only: Measurable disease as per RECIST v1.1 criteria (Note: Measurable disease is NOT required for Phase 1 Dose Escalation).
7. Eastern Cooperative Oncology Group (ECOG) ≤ 1.
8. Life expectancy ≥ 12 weeks.
9. No known contraindications to leukapheresis, cyclophosphamide, fludarabine, or steroids.
10. Baseline laboratory values as shown in the following table:

    Minimum Laboratory Values for Study Entry Laboratory Assessment Criteria White blood cell count > 4,000/mm3 Absolute neutrophil count (ANC) ≥ 1,500/mm3 Platelets ≥ 100,000/mm3 Hemoglobin ≥ 10 g/dL Total bilirubin ≤ 1.5 x upper limit of normal (ULN) Aspartate amino transferase (AST) ≤ 3 x ULN Alanine transaminase (ALT) ≤ 3 x ULN Creatinine clearance by Cockroft-Gault equation 60 mL/min Oxygen saturation ≥ 92% on room air Albumin ≥ 3 g/dL
11. Left ventricular ejection fraction ≥ 50%.
12. Seronegative for human immunodeficiency virus (HIV) by antigen/antibody (Ag/Ab) testing.
13. Seronegative for hepatitis B and/or hepatitis C virus.
14. Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test is required.
15. Agreement by women and men of childbearing potential to use an effective method of birth control or abstain from heterosexual activity through at least 3 months after the last dose of CHM-2101.

Exclusion Criteria:

1. Previous treatment with CDH17-targeted therapies.
2. Unresolved toxicities from prior therapy except for chronic toxicity no greater than Grade 1 and stable > 30 days (Note: alopecia of any grade is not exclusionary).
3. Uncontrolled seizure activity and/or known central nervous system (CNS) metastases.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent.
5. Uncontrolled Crohn's disease, ulcerative colitis, or other autoimmune or inflammatory disorders of the GI tract. "Uncontrolled" is defined as requiring hospitalization, corticosteroids, or chronic medication increase (dosage or frequency) within the previous 6 months.
6. Liver involvement ≥ 50%.
7. Active infection requiring oral or IV antibiotics.
8. Current diagnosis of pleural effusions, interstitial lung disease, or heart failure of New York Heart Association Classification of Heart Failure Class III or IV.
9. Ongoing treatment with systemic corticosteroid therapy at doses of prednisone ≥ 20 mg/day or equivalent (lower doses of corticosteroid therapy are allowed until 7 days prior to leukapheresis).
10. No prior malignancy within 5 years except for non-melanomatous skin cancer or cervical cancer treated with curative intent
11. Currently breastfeeding or planning to become pregnant within 9 months of study enrollment.
12. Any other clinically significant uncontrolled illness or other comorbid condition that would, in the investigator's judgment, contraindicate the participant's participation in the clinical study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | 28 Days
  Assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Rates and Grades of Cytokine Release Syndrome (CRS) | up to 15 years
  Assessed per American Society for Transplant and Cellular Therapy (ASTCT) consensus grading guideline
All other adverse events and toxicities | up to 15 years
  Assessed per NCI CTCAE v5.0
Objective Response Rate (ORR) | up to 15 years
  Assessed by RECIST v 1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 15 years
  Assessed as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response, and stable disease to a therapeutic intervention in clinical trials of anticancer agents.
Time to response (TTR) | up to 15 years
  Measured as the amount of time elapsed until drug response is achieved for the first time.
Duration of response (DOR) | up to 15 years
  Measured as the amount of time a patient responds to a treatment before disease progresses or the patient dies.
Progression-free survival (PFS) | up to 15 years
  Measured from the date of first infusion of CAR-T cells until the first date when progressive disease (PD) is objectively documented or death from any cause, whichever is earlier.
Overall survival (OS) | up to 15 years
  Measured from the date of first infusion of CAR-T cells until death.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Eads, MD, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No